CLINICAL TRIAL: NCT01964742
Title: Analysis of Host Genetic Factors in the Occurrence of Anemia and on the Virological Response to a Peg-interferon/Ribavirin Therapy in HIV-HCV Co-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-A00505-40; 2013-12 (Other: AP HM)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: HIV-HCV Co-infected Patients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV-HCV co-infected patients (Experimental)
  Interventions: Genetic: blood samples

INTERVENTIONS:
Genetic: blood samples

SUMMARY:
The treatment of HCV (hepatitis C virus) infection has made significant progress over the past decade with the therapy combining pegylated interferon (Peg-IFN) to ribavirin (RBV). The cure of HCV infection which consists to obtain a sustained virological response (SVR) (undetectable HCV RNA 24 weeks after end of treatment) is reached in more than 50% of patients infected with HCV. However, this rate is much lower, around 30 to 40% in HIV-HCV co-infected patients and sometimes can be less than 20% for patients infected with HCV genotype 1. Haemolytic anemia is a dose-limiting adverse effect which occurs frequently under RBV therapy. RBV-induced anemia represents the main cause of treatment discontinuation or dose reduction of RBV, thus limiting the chances of achieving a SVR. RBV has a large inter-individual pharmacokinetic variability and a relationship between the occurrence of anemia and RBV concentration was clearly demonstrated. However, other factors, including genetic factors, could be predictive of hematotoxicity and/or a better efficiency. In particular, IL-28B polymorphism analysis, in patients infected with HCV genotype 1, before starting antiviral therapy could predict the response to treatment (positive predictive value). The genetic polymorphism of inosine triphosphate pyrophosphatase (ITPA) is also strongly associated to a protective effect towards the RBV-induced-anemia. But most of these data are issued from studies performed in a Japanese HCV mono-infected population treated with Peg-IFN-RBV therapy for which there is no other causal variant that the rs1127354. Only few studies are reported in the literature in caucasian HIV-HCV co-infected patients. Moreover, data on RBV plasma exposure are very scarce in all these studies showing an impact of the ITPA polymorphism on the occurrence of anemia. In addition, others polymorphisms of SCL29A1/A2 and SCL28A2/A3 coding for RBV transporters, ENT (equilibrative nucleoside transporter) et CNT (concentrative nucleoside transporter) would be associated to either rapid virological response or anemia in HCV infected patients treated by Peg-IFN plus RBV. No study considering both polymorphisms of ITPA, IL-28B, SCL29A1/A2 and SCL28A2/A3 genes and RBV plasma exposure data has so far been conducted in HIV-HCV co-infected patients.

Thus, it would be interesting in a first time to assess the impact of the ITPA polymorphism on both the RBV plasma exposure and the protective effect towards RBV-induced anemia in HIV-HCV co-infected patients. This study could be helpful to the literature for possible further RBV dose adjustments according to ITPA activity.

Then, it would be relevant to further complete these data by assessing other genetic polymorphisms as IL-28B, SCL29A1/A2 and SCL28A2/A3 and thus evaluate the overall pharmacogenetic relationships towards RBV-induced anaemia and/or virological response to a Peg-IFN/RBV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Patients co-infected HIV-HCV (HCV serology and HCV positive CV before starting HCV treatment)
* Patients who have been treated with combination therapy Peg-IFN/RBV for at least 12 weeks and having at least a given plasma RBV available in the patient record
* Free Consent, informed and signed

Exclusion Criteria:

* Adult <18
* Mono-infection with HCV or HIV
* Co-infection with HBV (HBsAg +)
* Pregnant or lactating woman
* Not obtaining free and informed consent signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
blood samples | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France